CLINICAL TRIAL: NCT04719039
Title: The Effect of Restorative Yoga Self-Practice on Sleep Disturbance: A Pilot Randomized Controlled Trial
Brief Title: The Effect of Yoga Self-Practice on Sleep Disturbance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY014
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Yoga
Keywords: Insomnia; Yoga; Mindful breathing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Restorative Yoga intervention
  Interventions: Behavioral: Restorative Yoga Internvention
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive the intervention after the immediate post-treatment assessment

INTERVENTIONS:
Behavioral: Restorative Yoga Internvention — Participants in the intervention group will receive links to two 60-min videos per week for 8 consecutive weeks. Each video will include a yoga practice guided by a certified yoga instructor. The intervention group is required to perform the yoga practice at least two times per week. If preferred, they can do additional sessions with the videos and record their total hours of self-practice.
  Arms: Yoga Group

SUMMARY:
The study will examine the effect of Restorative Yoga self-practice on sleep disturbance in the Chinese adult population. Restorative Yoga is a relaxation-focused yoga style which includes a series of static stretching poses and mindful breathing. Existing literature has demonstrated that face-to-face yoga sessions of different types are effective in improving sleep disturbance and reducing the severity of insomnia. There were pilot studies conducted on the effect of yoga on cancer patients' sleep quality, but research that focuses on insomnia population is rare (Wang et al., 2020). In addition, there is very limited research on the effectiveness of self-practice without the presence of a yoga instructor. Given the social distancing policy under COVID-19 and the need to stay home, this study can shed light on whether self-practice at home can be an effective alternative to face-to-face yoga sessions.

DETAILED DESCRIPTION:
This study will be a pilot randomized controlled trial on the effectiveness of restorative yoga self-practice for sleep disturbance. Prior to all study procedures, online informed consent (with phone support) will be obtained from potential participants. Around 30 eligible participants will be randomly assigned to either the yoga group (intervention group) or the waitlist control group in a ratio of 1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. No deception is necessary.

Participants in the intervention group will receive links to two 60-min videos per week for 8 consecutive weeks. Each video will include a yoga practice guided by a certified yoga instructor. The intervention group is required to perform the yoga practice at least two times per week. If preferred, they can do additional sessions with the videos and record their total hours of self-practice. The waitlist control group will receive the video links subsequent to the 8-week study. The intervention group will complete a set of online questionnaires before the intervention commences, weekly during the intervention period, immediately after the intervention, and 4 weeks after the intervention. The waitlist control group will complete the same set of online questionnaires before the intervention commences and immediately after 8-week intervention period has ended.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18-59 years;
2. Cantonese language fluency;
3. A global Insomnia Severity Index (ISI) score of 10 or higher;
4. No yoga experience within the 6 months before the study; and
5. A willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

Participants were excluded if they

1. are pregnant;
2. are having unsafe conditions and are not recommended for restorative yoga by physicians;
3. have major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the yoga practice;
4. have insomnia due to specific medical conditions, side effects of medication intake or other sleep disorders; and
5. are shift workers.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, intervention period (8 weeks), immediate and 4-week post-intervention
  The PSQI-19 is a 19-item questionnaire used for measuring and identifying quality of sleep.
  It provides a measure of global sleep quality, including sleep latency, sleep duration, habitual sleep efficiency and sleep disturbances.
Change in Insomnia Severity Index (ISI) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Sleep Diary - Change in sleep-Onset latency (SOL) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  The standardized sleep diary records the length of time that it takes to accomplish the transition from full wakefulness to sleep on a daily basis.
Sleep Diary - Change in wake after sleep onset (WASO) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  The standardized sleep diary records the periods of wakefulness occurring after defined sleep onset on a daily basis, reflecting sleep fragmentation.
Sleep Diary - Change in total wake time (TWT) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  The standardized sleep diary records wake time to measure sleep disturbance.
Sleep Diary - Change in total sleep time (TST) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  The standardized sleep diary records wake time to measure sleep disturbance.
Sleep Diary - Change in sleep efficiency (SE) | Baseline, intervention period (8 weeks), immediately and 4-week post-intervention
  The Sleep efficiency is measured in percentage by dividing TST by total time in bed.

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS-14) | Baseline, immediately after the 8-week intervention, and 4-week post-intervention
  HADS is a 14-item self-rated questionnaire which consists of two 7-item subscales that measure the presence of anxiety and depression symptoms respectively. Each item is rated on a 4-point-scale (0-3) by the participant. The greater the score, the more psychologically distressed the respondent is.
Change in Multidimensional Fatigue Inventory (MFI-20) | Baseline, immediately after the 8-week intervention, and 4-week post-intervention
  The MFI-20 assesses the severity of fatigue covering the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.
Change in Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediately after the 8-week intervention, and 4-week post-intervention
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediately after the 8-week intervention, and 4-week post-intervention
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong